CLINICAL TRIAL: NCT01208493
Title: Dietary Protein in the Very-low-birth-weight Infant: Effects of the Level of Dietary Protein on Growth and Feeding Tolerance
Brief Title: Dietary Protein in the Very-low-birth-weight Infant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04.26.INF
Record Dates: First submitted 2010-09-22; First posted 2010-09-24 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2011-12

CONDITIONS: Prematurity
Keywords: prematurity; enteral feeding; proteins; formula
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high protein preterm infant formula (Experimental): preterm infant formula with high protein levels
  Interventions: Other: preterm infant formula with high protein levels
- control preterm formula (Active Comparator)
  Interventions: Other: preterm standard infant formula

INTERVENTIONS:
Other: preterm infant formula with high protein levels — minimum 3 weeks feeding until hospital discharge
  Arms: high protein preterm infant formula
Other: preterm standard infant formula — minimum 3 weeks feeding until hospital discharge
  Arms: control preterm formula

SUMMARY:
In this randomized study The investigators aim to compare the growth of very-low-birth-weight (VLBW) infants fed either a high protein or a standard protein preterm infant formula.

Babies will be fed the assigned formula between the time they achieve full enteral feeds and hospital discharge, for a minimum of 3 weeks. The weight gain (g/d) will be measured and compared between groups. Feeding tolerance, protein-energy status and body composition between the study groups will also be analysed.

After discharge, babies will be fed a post-discharge preterm infant formula (PDF) between hospital discharge and 3 m corrected age.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age <32 w, determined by maternal dates, fetal ultrasound, Dubowitz/Ballard examination or a combination thereof
* Birth weight ≤1500 g
* Tolerating an enteral intake of ≥100 ml/kg/d for ≥ 24 h
* Subject is anticipated to receive the study formula for ≥ 3 consecutive weeks after FEF have been achieved
* In infants fed human milk, formula is anticipated to provide 50% or more of total energy intake, calculated on a weekly basis and based on the assumption that human milk has an energy density of 67 kcal/dl
* Written informed consent has been obtained from the legal representative

Exclusion Criteria:

* Cardiac failure requiring fluid restriction with diuretic therapy for ≥ 3 consecutive days
* Peri-/intra-ventricular haemorrhage (grade 3-4) determined using cranial ultrasonography
* Renal disease: by symptoms (oliguria, anuria, proteinuria, hematuria) associated with an increased BUN and creatinine
* Sepsis: defined by symptoms requiring antibiotic therapy and confirmed by a positive blood culture
* Necrotizing Enterocolitis: defined by feeding intolerance associated with positive x-ray findings (pneumatosis intestinalis - Bell Stage 2; air in the biliary tract or free air in the peritoneum - Bell Stage 3)
* Hepatic dysfunction: defined by jaundice (direct bilirubin >1.0 mg/dl) which is associated with one or more abnormal liver function tests (AST, ALT or GGT)
* Lung disease, severe enough to require steroid therapy.
* Small size for gestational age (SGA) - body weight ≤ 5th percentile for that gestational age.
* Participation in another clinical trial that may affect outcomes of this study

Ages: 1 Day to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2007-09; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
comparison of weight gain between both study groups as a measure of safety | 3 weeks

SECONDARY OUTCOMES:
comparison of feeding tolerance and metabolic status between study groups as a measure of safety | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Cooke, MD, Principal Investigator — Department of Pediatrics St Louis University
Locations (4):
- Department of Pediatrics St Louis University, St Louis, Missouri, United States
- Service Universitaire de Néonatologie CHR de la Citadelle, Liège, Belgium
- Service de néonatologie Hôpital de la Croix Rousse, Lyon, France
- Department of Child Health Royal Victoria Infirmary, Newcastle upon Tyne, United Kingdom